CLINICAL TRIAL: NCT01171105
Title: A Phase I, Double-blind, Randomized, Placebo-controlled', Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral AZD5213 After Administration of Multiple Ascending Doses for 10 Days in Healthy Male and Non-fertile Female Volunteers
Brief Title: Study to Investigate Multiple Ascending Oral Doses of AZD5213 in Healthy Male and Non Fertile Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3030C00002
Record Dates: First submitted 2010-07-21; First posted 2010-07-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: AZD5213 Phase 1; Safety; tolerability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AZD5213 (dose escalating)
  Interventions: Drug: AZD5213
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo to AZD5213

INTERVENTIONS:
Drug: AZD5213 — oral solution, multiple ascending doses
  Arms: 1
Drug: Placebo to AZD5213
  Arms: 2

SUMMARY:
1. The main purpose of this study is to assess the safety and tolerability of AZD5213 after multiple oral doses.
2. Another purpose of this study is to evaluate the pharmacokinetics (also called PK - how the study drug enters and leaves your body and how your body acts on the study drug) of AZD5213 in your blood and urine.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-fertile female healthy volunteers aged 18-50 years and 65-80 years inclusive at day of enrollment with suitable veins for cannulation or repeated venipuncture.
* Male healthy volunteers should be willing to use barrier contraception during sexual intercourse, ie condoms, even if partner is using contraceptive method, from the first day of dosing until 3 months after the last dosing with AZD5213.
* Body weight of ≥50 to ≤100 Kg and Body Mass Index (BMI) ≥18 to ≤30 kg/m2.

Exclusion Criteria:

* History and presence of any clinically significant disease or disorder such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal and psychiatric/mental disorders.
* History or presence of gastrointestinal (including irritable bowel disease), hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs. Surgery on gastrointestinal tract.
* History of previous or ongoing psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Adverse events, vital signs, physical (including neurological) examinations, clinical laboratory variables, electrocardiograms, telemetry, sleep diary (temporal and qualitative aspects), and the Columbia-Suicide Severity Rating Scale | Up to 30 days screening period. Residential period will be 14 days. Follow up period will be 7 to 10 days after dose

SECONDARY OUTCOMES:
Multiple-dose PK and dose proportionality | Frequent timepoints within 48 hours of multiple dose day 1 and day 12.
Time to reach steady state | Frequent timepoints within 48 hours of multiple dose day 1 and day 12.
Degree of accumulation and time dependancy of orally-administered AZD5213 | Frequent timepoints within 48 hours of multiple dose day 1 and day 12.

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles, 6700 W. 115th Street, Overland Park, KS 66211
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: D3030C00002 Clinical Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1313&filename=D3030C00002_Clinical_Study_Report_Synopsis.pdf